CLINICAL TRIAL: NCT00778869
Title: Whole Human Genome Oligo Microarray Analysis of the Peripheral Blood Mononuclear Cells of Patients With Ankylosing Spondylitis During Infliximab Treatment Compared to Healthy Controls
Brief Title: Analysis of the Peripheral Blood Mononuclear Cells of Patients With Ankylosing Spondylitis During Infliximab Treatment (Study P04465)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04465
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remicade (Experimental): Remicade will be given at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54.
  Interventions: Biological: Remicade

INTERVENTIONS:
Biological: Remicade — Remicade will be given at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54.
  Other Names: Infliximab; SCH 215596

SUMMARY:
This is an open-label, controlled sub-study to the parent protocol (P04041, NCT00779935) to examine the expression profile of genes in patients in the active stage of ankylosing spondylitis (AS) compared to the healthy population as control, moreover to examine the changes in expression profile during anti-tumor necrosis factor (TNF)-alpha treatment (Remicade).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis proven by appropriate diagnostic methods (according to New York criteria).
* Refractory disease defined by failure of at least 2 non-steroidal anti-inflammatory drugs (NSAIDs) during a 3-month period and failure of sulfasalazine in subjects with associated peripheral arthritis.
* Active disease defined by:

  * sustained bath ankylosing spondylitis disease activity index (BASDAI) of at least 40 on a 0-100 scale and
  * expert opinion based on clinical features.
* Age between 18 and 70 years.
* Subjects using NSAIDs and/or sulfasalazine must have been on a stable dose for at least 4 weeks prior to study initiation, and may continue medication during the treatment period, but the dose must not be increased above the baseline.
* Subjects must be capable to demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Men and women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (eg, hormonal contraceptive, medically prescribed intrauterine device (IUD), condom in combination with spermicide) or be surgically sterilized (eg, hysterectomy or tubal ligation).
* Subjects must understand and be able to adhere to the dosing and visit schedules.

Exclusion Criteria:

* Subject with moderate or severe heart failure (New York Heart Association (NYHA) class III/IV).
* Remicade must not be given to subjects with a history of hypersensitivity to infliximab, to other murine proteins, or to any of the excipients.
* Subjects with pre-existing or recent onset of central nervous system demyelinating disorders.
* Age <18 or >70 years.
* Pregnant women, nursing mothers.
* Subjects who are incapacitated, largely or wholly bedridden or confined to a wheelchair, and who have little or no ability for self-care.
* Subjects who have any current systemic inflammatory condition with signs and symptoms that might confound the evaluations of benefit from infliximab therapy.
* Prior administration of infliximab or any other therapeutic agent targeted at reducing tumor necrosis factor (TNF) (eg, Etanercept, pentoxifylline, thalidomide or anti-CD4+ antibody).
* Current treatment with systemic corticosteroid.
* Treatment with any investigational drug within the previous 3 months.
* History of known allergies to murine proteins.
* Subjects having active or inactive tuberculosis (TB). All subjects must be evaluated for both active and inactive ('latent') TB. This evaluation should include a detailed medical history with personal history of TB or possible previous contact with TB and previous and/or current immunosuppressive therapy. Appropriate screening tests (ie, tuberculin skin test and chest x-ray) should be performed in all subjects.
* Serious infection, such as sepsis, abscesses, hepatitis, pneumonia, pyelonephritis in the previous 3 months. Less serious infections in the previous 3 months, such as acute respiratory tract infection (colds) or uncomplicated urinary tract infection need not be considered exclusions at the discretion of the treating physician.
* History of opportunistic infections such as herpes zoster within 2 months of study initiation. Evidence of active cytomegalovirus (CMV), active pneumocystis carinii, drug resistant atypical mycobacterium, etc.
* Documented human immunodeficiency virus (HIV) infection.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* Any currently known malignancy or pre-malignant lesions or any history of malignancy within the past 5 years (except non-melanoma skin cancer and surgically cured cervical cancer).
* Subjects with alcoholism, alcoholic liver disease, or other chronic liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Remicade: Remicade will be given as an intravenous infusion at a dose of 5 mg/kg at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54.
Period: Overall Study
Arm/Group | Remicade
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Remicade
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Genes Which Were Differentially Expressed
Description: Differentially expressed genes were described as those which were at least 1.5 times up- or down-regulated and statistically different at a significance level of 0.05 using a paired t-test comparing 10 ankylosing spondylitis (AS) participants during tumor necrosis factor (TNF) alpha treatment (Remicade) with 10 matched controls. Control samples were previously obtained and not specifically collected for this study.
Time Frame: 14 weeks
Measure: Number; unit: Number of genes
Groups:
- Remicade: Remicade will be given as an intravenous infusion at a dose of 5 mg/kg at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54 in participants with AS.
Arm/Group | Remicade
Number analyzed (Participants) | 10
Number of genes
  Number of Genes | 54675
  Number of Genes Up/Down Regulated | 890
  Number of Genes Highly Expressed | 701
Statistical Analysis 1: Comparison: Remicade; Test type: Superiority or Other; p < 0.05, Student t-test

ADVERSE EVENTS:
Description: Non-serious adverse events and serious adverse events were not required to be captured as part of the study database. They were captured in the parent protocol (P04041). Therefore, none were collected, and the number of participants at risk is zero.
Arm/Group | Remicade
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator (PI) agrees not to publish or publicly present any interim results of study without prior written consent of sponsor. PI further agrees to provide 30 days written notice to sponsor prior to submission for publication or presentation to permit sponsor to review copies of abstracts or manuscripts for publication including without limitation slides and texts of oral or other public presentations and text of any transmission through any electronic media which report results.